CLINICAL TRIAL: NCT06502054
Title: Being a Parent with an Autism Spectrum Disorder: Strengths, Challenges and Adaptation of a Mentalization-based Parenting Program
Brief Title: Parenting with an Autism Spectrum Disorder
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Johannes Boettcher, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: LPEK-0765
Record Dates: First submitted 2024-07-05; First posted 2024-07-15 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Parenthood; Autism Spectrum Disorder; Preschool children
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Autistic parents: Parents who fulfill the main diagnosis of ASD, which includes atypical autism (ICD-10: F84.1) and Asperger syndrome (ICD-10: F84.5), who are ≥ 18 years old and have a child aged 0 to 6 years are included.
- Non-autistic parents: Parents are included who do not have a lifetime main diagnosis of a psychiatric illness (ICD-10-GM-2016: F10 - F69), who are ≥ 18 years old and have a child aged 0 to 6 years.

SUMMARY:
In many individuals, Autism Spectrum Disorder (ASD) is recognized and diagnosed late in adolescence or even in adulthood, despite the presence of long-standing impairments and distress. One area that has received little attention so far is research and interventions in clinical practice that relate to the experienced realities of parenthood for autistic adults or offer support in this context. The few existing research findings in this field suggest that parents with ASD might face specific challenges. At the same time, there is a lack of empirical research on the experiences autistic adults have with parenthood, whether they perceive a need for specific support services, and, if so, what those services should look like. To fill this research gap, this study aims to examine the mental health, needs, and strengths of parents with ASD. Particular focus will be given to parental stress and difficulties in the areas of mentalization and emotion regulation, which can increase the risk of psychological comorbidities. Using a mixed-methods approach, the study will investigate to what extent an already established parenting program or an adaptation thereof might be suitable to address the specific requirements of autistic parents and enhance their parenting skills.

ELIGIBILITY:
In- and exclusion criteria for the study population:

Inclusion Criteria:

* Parents who fulfill the main diagnosis of ASD, including atypical autism (ICD-10: F84.1) and Asperger syndrome (ICD-10: F84.5)
* Age ≥ 18 years
* Have a child aged 0 to 6 years

Exclusion Criteria:

* Below-average general cognitive ability (according to clinical impression)
* Lack of German language skills
* Severe visual or hearing impairment (uncorrected)
* Serious neurological and psychiatric illnesses (e.g., epilepsy, psychoses)
* Acute suicidal tendencies (according to clinical findings)

Eligibility Criteria for the Control Group

Inclusion Criteria:

* Parents without a lifetime main diagnosis of a psychiatric illness (ICD-10-GM-2016: F10 - F69)
* Age ≥ 18 years
* Have a child aged 0 to 6 years
* Matched to the study group in terms of age and gender

Exclusion Criteria:

* Above-mentioned psychiatric diagnoses
* Below-average general cognitive ability
* Lack of German language skills
* Severe impairment of vision or hearing (not corrected)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents who fulfill the main diagnosis of ASD, who are ≥ 18 years old and have a child aged 0 to 6 years.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Mentalization | Baseline assessment
  The Mentalization Scale (MentS) is a 28-item instrument for measuring mentalization in three aspects: self-related, other-related, and motivation to mentalize. The total score for the MentS ranges from 28 to 140, with higher scores indicating a higher overall ability to mentalize. Higher scores in the subscales and total score indicate a higher ability to mentalize.

SECONDARY OUTCOMES:
Autistic Traits | Baseline assessment
  The Autism Spectrum Quotient-10 (AQ-10) is a shortened self-report questionnaire developed to measure autistic traits in adults. The instrument is a brief version of the Autism Spectrum Quotient and consists of 10 items that can be used as a screening tool. The total score for the Autism Spectrum Quotient-10 ranges from 0 to 10, with higher scores indicating a higher presence of autistic traits.
Parental Quality of Life | Baseline assessment
  The Short-Form Health Survey - 12 (SF-12) is a screening instrument for assessing health-related quality of life. The SF-12 includes the Physical Component Summary score representing General Health Perception, Physical Functioning, Role Physical, and Bodily Pain, and the Mental Component Summary score reflecting Emotional Role Functioning, Mental Health, Vitality, and Social Functioning. Scores for the SF-12 typically range from 0 to 100 for each summary component, with higher scores indicating better health-related quality of life.
Parental mental health | Baseline assessment
  The Brief Symptom Inventory-18 (BSI-18) is a shortened version of the Symptom Checklist 90, consisting of 18 items. The BSI-18 short form is a cost-effective, reliable, and valid self-report measure that is increasingly internationally recognized. It comprises 6 items each assessing the syndromes of somatization, depression, and anxiety. Scores for the BSI-18 range from 0 to 72, with higher scores indicating greater symptom severity.
Children mental health | Baseline assessment
  The Strengths and Difficulties Questionnaire (SDQ) is one of the most commonly used measures for assessing the mental health of children and adolescents from both self and parent perspectives. The SDQ assesses mental health issues and resources in children and adolescents aged 2 to 17 years with five items each across five subscales: conduct problems, emotional symptoms, hyperactivity, peer problems, and prosocial behavior. Scores for each subscale range from 0 to 10, and the total difficulties score ranges from 0 to 40. Higher scores on the conduct problems, emotional symptoms, hyperactivity, and peer problems subscales indicate greater difficulties, while higher scores on the prosocial behavior subscale indicate greater strengths.

OTHER OUTCOMES:
Emotion regulation | Baseline assessment
  The Difficulties in Emotion Regulation Scale - Short Form (DERS-SF) is an 18-item questionnaire designed to assess emotion regulation difficulties in adults. The measurement covers four dimensions of emotion regulation: awareness and understanding of emotions; acceptance of emotions; the ability to engage in goal-directed behavior and refrain from impulsive behavior when experiencing negative emotions; and access to perceived effective emotion regulation strategies. Scores for the DERS-SF range from 18 to 90, with higher scores indicating greater difficulties in emotion regulation.
Parental stress | Baseline assessment
  The Parental Stress Inventory (Eltern-Belastungs-Inventar; EBI) is an instrument for assessing parental stress. The Parental Stress Inventory comprises a total of 48 items. It provides indications of whether parents are impaired in their tasks of parenting, caring, and providing for their child due to increased stress, thus necessitating support or intervention measures for the family. Scores for the Parental Stress Inventory range from 48 to 240, with higher scores indicating greater parental stress.
Self-efficacy in parenting | Baseline assessment
  The Parenting Self-Efficacy Questionnaire (Fragebogen zur Selbstwirksamkeit in der Erziehung; FSW) is a 9-item questionnaire designed to assess parenting self-efficacy. Scores for the Parenting Self-Efficacy Questionnaire range from 9 to 45, with higher scores indicating greater self-efficacy in parenting.
Mentalization II | Baseline assessment
  The Certainty About Mental States Questionnaire (CAMSQ) is a self-assessment instrument for measuring the perceived ability to understand mental states of oneself and others (i.e., mentalizing). The CAMSQ consists of 20 items answered on a seven-point response scale. Scores for the Certainty About Mental States Questionnaire range from 20 to 140, with higher scores indicating a greater perceived ability to understand mental states.
Mentalization III | Baseline assessment
  The Parental Reflective Functioning Questionnaire (PRFQ) will be used to assess Parental Reflective Functioning (PRF) as a multidimensional construct. The PRFQ consists of 18 items rated on a 7-point Likert scale. Scores for the Parental Reflective Functioning Questionnaire range from 18 to 126, with higher scores indicating greater parental reflective functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No